CLINICAL TRIAL: NCT00692198
Title: Effectiveness of Long-term Oxygen Therapy in Treating People With Chronic Obstructive Pulmonary Disease With Moderate Desaturation
Brief Title: Long-term Oxygen Treatment Trial
Acronym: LOTT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: Centers for Medicare and Medicaid Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 583; N01HR76197-12-0-3 (NIH)
Record Dates: First submitted 2008-06-04; First posted 2008-06-06 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2017-05-10 (Actual); Status verified 2016-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Supplemental oxygen therapy (Experimental): Participants will receive treatment with supplemental oxygen therapy.
  Interventions: Drug: Supplemental oxygen therapy
- No supplemental oxygen therapy (No Intervention): Participants will receive no supplemental oxygen therapy, unless the participant becomes severely hypoxemic at rest (e.g., meets conventional Medicare criteria for 24-hour supplemental oxygen due to severe hypoxemia at rest).

INTERVENTIONS:
Drug: Supplemental oxygen therapy — Oxygen dose at rest and during sleep will be 2 L/min via nasal cannula. The oxygen dose used while walking will be individually prescribed and will be sufficient to maintain oxygen saturation at 90% or above for at least 2 minutes while walking. Participants who have low blood oxygen levels at rest will be instructed to use oxygen 24 hours per day. Participants who have normal resting blood oxygen levels, but low or very low blood oxygen levels during exercise, will be instructed to use oxygen during physical activity and sleep.
  Arms: Supplemental oxygen therapy

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a serious respiratory disease in which the airways in the lungs are partially blocked, resulting in symptoms of chest tightness, coughing, and difficulty breathing. Currently, there are many available treatments for managing COPD symptoms and improving quality of life, including medications, lifestyle changes, oxygen therapy, and pulmonary rehabilitation. For people with severe COPD that is characterized by very low blood oxygen levels at rest, long term oxygen therapy can help to prolong life and promote feelings of well-being. However, the effectiveness of supplemental oxygen therapy for people with COPD that is characterized by only moderately low blood oxygen levels at rest or normal blood oxygen at rest and desaturation on exercise is not known. This study will evaluate the effectiveness of supplemental oxygen therapy in treating people with COPD who have moderately low blood oxygen levels at rest or who have normal blood oxygen levels at rest, but have low or very low blood oxygen levels during exercise.

DETAILED DESCRIPTION:
COPD is the fourth leading cause of death in the United States, with more than 12 million people currently diagnosed with the disease. Risk factors for COPD include smoking, environmental exposure to lung irritants, and genetic predisposition. People with COPD often experience symptoms of chronic cough, shortness of breath, excess mucus production, and wheezing. In COPD, the airways in the lungs are chronically obstructed, and if left untreated, this obstruction can cause significant damage to the lungs and lasting disability. The quality of life of a person with COPD decreases as the disease progresses, making treating and managing COPD in the moderate stages important. Long-term oxygen therapy has been shown to help people with severe COPD that is characterized by very low blood oxygen levels at rest to live longer and healthier lives. This study will determine whether supplemental oxygen therapy is helpful for people with COPD that is characterized by moderately low blood oxygen levels at rest or normal oxygen levels at rest and low or very low levels during exercise.

Participation in this study will last at least one year and up to 7 years. Potential participants will first undergo a screening visit that will include questionnaires, a breathing test, measurements of resting and walking blood oxygen levels, a brief physical exam, and a blood draw. Eligible participants will then return for a second screening visit, during which they will complete more questionnaires. At the end of the second visit, eligible participants will be assigned randomly to supplemental oxygen therapy or no oxygen therapy.

Participants assigned to supplemental oxygen therapy will receive stationary and portable oxygen systems. Shortly after receiving the portable oxygen system, participants will return for a 1-hour visit to determine how much oxygen to use while walking and to learn how to use the equipment. Participants who have low blood oxygen levels during rest will be instructed to use supplemental oxygen 24 hours per day. Patients with normal resting blood oxygen levels, but low or very low blood oxygen levels during exercise will be instructed to use it during physical activity and sleep. Throughout the treatment period, participants will be asked to keep records of the number of oxygen tanks emptied or pounds of oxygen delivered, meter readings, and changes in equipment. Study officials will contact participants weekly for the first month, monthly for the next 5 months, and then every 2 months until the Year 1 study visit. Participants will also complete a form about their oxygen equipment and usage every 2 months. Participants assigned to receive no oxygen treatment will be contacted 1 week after study group assignment for a check-up.

All participants will return for study visits once a year for up to 7 years. At each of these visits, participants will complete some of the same tests and questionnaires from the screening visit. At the Year 1 visit, participants will also undergo a blood draw. Both treatment groups will receive two phone calls each year to check on status and use of oxygen. Participants in both groups will be asked to complete a quality of life questionnaire by mail at 4 months and 16 months. Participants will also sign a release of medical records form each year and will have their Medicare claims collected for the time they are in the study.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 40 years
* COPD
* Dyspnea, determined by Modified Medical Research Council (MMRC) scale of at least 1
* Dyspnea and lung disease process dominated by COPD in judgment of the study physician
* Participant must meet one of the following:

  * Post-bronchodilator forced expiratory volume in 1 second (FEV1) percent less than or equal to 70% predicted
  * Post-bronchodilator forced expiratory volume in 1 second (FEV1) percent >70% predicted and LOTT study physician determines that there is radiologic evidence of emphysema
* Post-bronchodilator FEV1/forced vital capacity (FVC) less then 0.70
* Participant must meet either of the following oxygen saturation criteria:

  * Oxygen saturation of at least 89% and no greater than 93% after sitting quietly on room air, without hyperventilation and without pursed lips breathing during oximetry
  * Resting oxygen saturation 94% or greater and desaturation during exercise defined as saturation below 90% for at least 10 seconds during the 6 minute walk test
* If participant is on supplemental oxygen at the start of screening, all of the following must be met prior to randomization:

  * Participant agrees to stop using oxygen if randomized to no oxygen
  * Participant's physician agrees in writing to rescind order for oxygen if participant is randomized to no oxygen
  * Participant must report not using oxygen on the day of randomization and must report not using oxygen for the 4 calendar days prior to randomization
  * Satisfactory resolution of logistics of continuation with same oxygen company with waiver of cost sharing obligations or switch to new company that will waive cost sharing obligations if participant is randomized to oxygen
* At least 10 pack-years of tobacco cigarette smoking before study entry
* Agreement not to smoke while using supplemental oxygen
* Medicare beneficiary with both Part A and Part B coverage or insurance OR personally willing to cover costs typically covered by Medicare
* Approval of study physician for randomization to either treatment group
* Completion of all required prerandomization assessments within 60 days of initiating study entry
* Randomization within 60 days of initiating eligibility evaluation
* Consent

Exclusion Criteria:

* Less than 30 days post treatment for acute exacerbation of COPD as of initiating eligibility evaluation (less than 30 days from last dose of antibiotics or since a new or increased dose of systemic corticosteroids was initiated); chronic use of systemic corticosteroids while health is stable is not exclusionary
* COPD exacerbation requiring antibiotics, new or increased dose of systemic corticosteroids, or oxygen treatment after screening starts and prior to randomization (chronic use of corticosteroids while health is stable is not exclusionary)
* Less than 30 days post discharge from an acute care hospital after acute care hospitalization for COPD or other condition, as of initiating eligibility evaluation (participant may be in a rehab hospital at time of screening)
* New prescription of supplemental oxygen after screening starts and before randomization
* Thoracotomy, sternotomy, major cardiopulmonary intervention (e.g., lung resection, open heart surgery, etc.), or other procedure in the 6 months before study entry likely to cause instability of pulmonary status
* Non-COPD lung disease that affects oxygenation or survival
* Epworth Sleepiness Scale score greater than 15
* Desaturation below 80% for at least 1 minute during the 6-minute walk test
* Disease or condition expected to cause death, inability to perform procedures for the trial, or inability to comply with therapy within 6 months of random assignment, as judged by the study physician
* Participation in another intervention study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 738 (Actual)
Dates: Start 2009-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William C. Bailey, MD, Study Chair — University of Alabama at Birmingham Lung Health Center
Locations (39):
- United States (39):
  - Birmingham VA Medical Center, Birmingham, Alabama
  - University of Alabama, Birmingham, Alabama
  - City of Hope National Medical Center, Duarte, California
  - Loma Linda VA Medical Center, Loma Linda, California
  - Los Angeles Biomedical Research Institute at Harbor-UCLA Medical Center, Los Angeles, California
  - UCSD Medical Center, San Diego, California
  - Denver Health and Hospital Authority, Denver, Colorado
  - National Jewish Medical and Research Center, Denver, Colorado
  - North Florida/South Georgia VA, Gainseville, Florida
  - Central Florida Pulmonary Group, Orlando, Florida
  - Weston Florida Cleveland Clinic, Weston, Florida
  - University of Illinois at Chicago, Chicago, Illinois
  - Suburban Lung Associates, Elk Grove Village, Illinois
  - Louisiana State University Health Sciences Center, New Orleans, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Boston VA Medical Center, West Roxbury, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Beaumont Hospital, Royal Oak, Michigan
  - Washington University, St Louis, Missouri
  - Pulmonary Consultants Inc./Christian Hospital, St Louis, Missouri
  - Buffalo VAMC, Buffalo, New York
  - Crouse Medical Practice, Syracuse, New York
  - Duke University, Durham, North Carolina
  - Cincinnati VA Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Kaiser Foundation Hospitals, Portland, Oregon
  - Geisinger Institute, Danville, Pennsylvania
  - Institute for Respiratory and Sleep Medicine, Langhorne, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Respiratory Specialists, Wyomissing, Pennsylvania
  - University of Texas at San Antonio, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
  - Harborview Medical Center, Seattle, Washington
  - University of Washington, Seattle, Washington
  - Puget Sound VA Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Datasets and associated documentation will be deposited with the National Heart, Lung, and Blood Institute Biologic Specimen and Data Repository Information Coordinating Center (NHLBI BioLINCC) repository once the contract ends, currently scheduled for May 2017. Data will be deidentified per BioLINCC requirements; datasets will include baseline and follow-up data collected during the trial. The BioLINCC Repository website includes instructions regarding accessing data on deposit in their repository.

REFERENCES:
- [Result] Long-Term Oxygen Treatment Trial Research Group; Albert RK, Au DH, Blackford AL, Casaburi R, Cooper JA Jr, Criner GJ, Diaz P, Fuhlbrigge AL, Gay SE, Kanner RE, MacIntyre N, Martinez FJ, Panos RJ, Piantadosi S, Sciurba F, Shade D, Stibolt T, Stoller JK, Wise R, Yusen RD, Tonascia J, Sternberg AL, Bailey W. A Randomized Trial of Long-Term Oxygen for COPD with Moderate Desaturation. N Engl J Med. 2016 Oct 27;375(17):1617-1627. doi: 10.1056/NEJMoa1604344. PMID 27783918
- [Derived] Moy ML, Harrington KF, Sternberg AL, Krishnan JA, Albert RK, Au DH, Casaburi R, Criner GJ, Diaz P, Kanner RE, Panos RJ, Stibolt T, Stoller JK, Tonascia J, Yusen RD, Tan AM, Fuhlbrigge AL; LOTT Research Group. Characteristics at the time of oxygen initiation associated with its adherence: Findings from the COPD Long-term Oxygen Treatment Trial. Respir Med. 2019 Mar;149:52-58. doi: 10.1016/j.rmed.2019.02.004. Epub 2019 Feb 13. PMID 30803886
- [Derived] Yusen RD, Criner GJ, Sternberg AL, Au DH, Fuhlbrigge AL, Albert RK, Casaburi R, Stoller JK, Harrington KF, Cooper JAD Jr, Diaz P, Gay S, Kanner R, MacIntyre N, Martinez FJ, Piantadosi S, Sciurba F, Shade D, Stibolt T, Tonascia J, Wise R, Bailey WC; LOTT Research Group *; LOTT Research Group. The Long-Term Oxygen Treatment Trial for Chronic Obstructive Pulmonary Disease: Rationale, Design, and Lessons Learned. Ann Am Thorac Soc. 2018 Jan;15(1):89-101. doi: 10.1513/AnnalsATS.201705-374SD. PMID 29087741
- [Derived] Stoller JK, Aboussouan LS, Kanner RE, Wilson LA, Diaz P, Wise R; LOTT Research Group. Characteristics of Alpha-1 Antitrypsin-Deficient Individuals in the Long-term Oxygen Treatment Trial and Comparison with Other Subjects with Chronic Obstructive Pulmonary Disease. Ann Am Thorac Soc. 2015 Dec;12(12):1796-804. doi: 10.1513/AnnalsATS.201506-389OC. PMID 26653189
- See also: Click here for more information about the Long-term Oxygen Treatment Trial — https://jhuccs1.us/lott/

RESULTS

PARTICIPANT FLOW:
Groups:
- Supplemental Oxygen Therapy (LTOT): Participants will receive treatment with supplemental oxygen therapy.
  Supplemental oxygen therapy: Oxygen dose at rest and during sleep will be 2 L/min via nasal cannula. The oxygen dose used while walking will be individually prescribed and will be sufficient to maintain oxygen saturation at 90% or above for at least 2 minutes while walking. Participants who have low blood oxygen levels at rest will be instructed to use oxygen 24 hours per day. Participants who have normal resting blood oxygen levels, but low or very low blood oxygen levels during exercise, will be instructed to use oxygen during physical activity and sleep.
- No Supplemental Oxygen Therapy (No LTOT): Participants will receive no supplemental oxygen therapy, unless the participant becomes severely hypoxemic at rest (e.g., meets conventional Medicare criteria for 24-hour supplemental oxygen due to severe hypoxemia at rest) or during exercise (SpO2 below 80% for at least 1 minute during 6 minute walk).
Period: Overall Study
Arm/Group | Supplemental Oxygen Therapy (LTOT) | No Supplemental Oxygen Therapy (No LTOT)
Started | 368 | 370
Completed | 368 | 370
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Supplemental Oxygen Therapy | No Supplemental Oxygen Therapy | Total
Number analyzed (Participants) | 368 | 370 | 738
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.3 (7.5) | 69.3 (7.4) | 68.8 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 94 | 196
  Male | 266 | 276 | 542
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 4 | 14
  Not Hispanic or Latino | 358 | 366 | 724
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: African American only | 46 | 34 | 80
  Race: Caucasian only | 299 | 322 | 621
  Race: Other | 23 | 14 | 37
Region of Enrollment [Number; unit: participants]
  United States | 368 | 370 | 738
Medicare coverage [Count of Participants; unit: Participants] | 268 | 273 | 541
Current tobacco-cigarette smoker [Count of Participants; unit: Participants] | 110 | 92 | 202
Quality of Well-Being Scale mean daily score [Mean (Standard Deviation); unit: units on a scale] — The Quality of Well Being questionnaire measures health related quality of life and is comprised of of 79 self reported items. The total daily score ranges from 0 to 1, with higher score indicating higher quality of life.
  units on a scale | 0.56 (0.13) | 0.56 (0.13) | 0.56 (0.13)
St George's Respiratory Questionnaire total score [Mean (Standard Deviation); unit: units on a scale] — The St George's Respiratory Questionnaire measures the impact of chest disease on daily life and well-being and is comprised of 51 items. The total score ranges from 0 to 100 with lower scores indicating better functioning.
  units on a scale | 49.8 (18.7) | 50.2 (17.1) | 50.0 (17.9)
Oxygen desaturation type qualifying patient for enrollment [Count of Participants; unit: Participants]
  Resting desaturation only | 73 | 60 | 133
  Exercise desaturation only | 148 | 171 | 319
  Resting and exercise | 147 | 139 | 286
SpO2 at rest while breathing ambient air [Mean (Standard Deviation); unit: SpO2 (percent saturation)] | 93.3 (2.1) | 93.5 (1.9) | 93.4 (2.0)
Nadir SpO2 during 6-min walk while breathing ambient air [Count of Participants; unit: Participants]
  Less than 86% | 86 | 85 | 171
  86% through 88% | 105 | 103 | 208
  Greater than 88% | 101 | 102 | 203
  Unknown | 76 | 80 | 156

OUTCOME MEASURES:

1. Primary Outcome: Death or Hospitalization, Whichever Occurs First
Description: The primary outcome event is death or hospitalization, whichever occurs first. The difference between treatment groups on the primary outcome was assessed with a time-to-event analysis by calculation of the between group hazard ratio for the primary composite outcome; the statistical significance of the hazard ratio was determined from the log rank test. The uncertainty in the hazard ratio is expressed in the 95% confidence interval on the hazard ratio.
Time Frame: Through study completion. Median follow-up was 18.4 months.
Measure: Number; unit: Composite events/100 person-years
Groups:
- No Supplemental Oxygen Therapy: Participants will receive no supplemental oxygen therapy, unless the participant becomes severely hypoxemic at rest (e.g., meets conventional Medicare criteria for 24-hour supplemental oxygen due to severe hypoxemia at rest) or during exercise (SpO2 below 80% for at least 1 minute during 6 minute walk).
Arm/Group | Supplemental Oxygen Therapy | No Supplemental Oxygen Therapy
Number analyzed (Participants) | 368 | 370
Composite events/100 person-years | 34.2 | 36.4
Statistical Analysis 1: Comparison: Supplemental Oxygen Therapy vs No Supplemental Oxygen Therapy; Test type: Superiority or Other; p = 0.52, Log Rank; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.79 to 1.12]

2. Secondary Outcome: Death
Description: The difference between treatment groups in mortality is assessed with a time-to-event analysis by calculation of the between group hazard ratio for death; the statistical significance of the hazard ratio was determined from the log rank test. The uncertainty in the hazard ratio is expressed in the 95% confidence interval on the hazard ratio.
Time Frame: Through study completion. Median follow-up was 41.5 months.
Measure: Number; unit: Deaths/100 person-years
Arm/Group | Supplemental Oxygen Therapy | No Supplemental Oxygen Therapy
Number analyzed (Participants) | 368 | 370
Deaths/100 person-years | 5.2 | 5.7
Statistical Analysis 1: Comparison: Supplemental Oxygen Therapy vs No Supplemental Oxygen Therapy; Test type: Superiority or Other; p = 0.53, Log Rank; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.64 to 1.25] — Hazard ratio, LTOT vs No LTOT

3. Secondary Outcome: Health Care Utilization
Description: Health care utilization is measured by the rate of all hospitalizations.
Time Frame: Through study completion. Median follow-up was 18.4 months.
Measure: Number; unit: Hospitalizations per 100 person-years
Arm/Group | Supplemental Oxygen Therapy | No Supplemental Oxygen Therapy
Number analyzed (Participants) | 368 | 370
Hospitalizations per 100 person-years | 56.9 | 56.2
Statistical Analysis 1: Comparison: Supplemental Oxygen Therapy vs No Supplemental Oxygen Therapy; Test type: Superiority or Other; p = 0.81, Fisher Exact; Rate ratio = 1.01, 95% CI 2-sided [0.91 to 1.13] — Rate ratio, LTOT vs No LTOT

4. Secondary Outcome: Adherence
Description: Adherence is measured by self-reported hours of home oxygen per day
Time Frame: Through study completion. Median follow-up was 18.4 months.
Population: Patients providing at least 1 self-report are included.
Measure: Mean (Standard Deviation); unit: hours per day of supplemental oxygen
Arm/Group | Supplemental Oxygen Therapy | No Supplemental Oxygen Therapy
Number analyzed (Participants) | 368 | 363
hours per day of supplemental oxygen | 13.6 (6.1) | 1.8 (3.9)

5. Secondary Outcome: COPD Exacerbation
Description: Rate of all COPD exacerbations
Time Frame: Through study completion. Median follow-up was 11.4 months
Measure: Number; unit: COPD exacerbations per 100 person-years
Arm/Group | Supplemental Oxygen Therapy | No Supplemental Oxygen Therapy
Number analyzed (Participants) | 368 | 370
COPD exacerbations per 100 person-years | 73.1 | 67.7
Statistical Analysis 1: Comparison: Supplemental Oxygen Therapy vs No Supplemental Oxygen Therapy; Test type: Superiority or Other; p = 0.12, Fisher Exact; Rate ratio = 1.08, 95% CI 2-sided [0.98 to 1.19] — Rate ratio, LTOT vs No LTOT

6. Secondary Outcome: Preference-weighted Health-related Quality of Life
Description: Preference-weighted health-related quality of life is measured by change in the Quality of Well-being Scale total daily score, follow-up value minus baseline value. The total daily score ranges from 0 to 1 with higher score indicating more better quality of life. Death is scored 0. Greater change, follow-up minus baseline, indicates improvement in quality of life compared to baseline. Change scores may range from -1 to +1.
Time Frame: Baseline to 1 year
Population: Participants with both the baseline and 1 year values were included
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Supplemental Oxygen Therapy | No Supplemental Oxygen Therapy
Number analyzed (Participants) | 341 | 312
units on a scale | -0.04 (0.24) | -0.04 (0.14)
Statistical Analysis 1: Comparison: Supplemental Oxygen Therapy vs No Supplemental Oxygen Therapy; Test type: Superiority or Other; p = 0.73, t-test, 2 sided

7. Secondary Outcome: Disease-specific Quality of Life
Description: Disease-specific quality of life is measured by the change in the St George's Respiratory Questionnaire total score, follow-up value minus baseline value. The total score ranges from 0 to 100 with lower score indicating fewer respiratory symptoms. Change in score, follow-up minus baseline may range from -100 to +100, with lower values indicating improvement in disease-specific quality of life.
Time Frame: Baseline to 1 year
Population: Participants with both the baseline and 1 year values are included
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Supplemental Oxygen Therapy | No Supplemental Oxygen Therapy
Number analyzed (Participants) | 331 | 299
units on a scale | -1.1 (13.5) | 0.6 (12.7)
Statistical Analysis 1: Comparison: Supplemental Oxygen Therapy vs No Supplemental Oxygen Therapy; Test type: Superiority or Other; p = 0.21, t-test, 2 sided

8. Secondary Outcome: General Quality of Life
Description: General quality of life is measured by the change in the physical component summary subscale of the SF-36 quality of life questionnaire, follow-up value minus baseline value. The physical component summary subscale score ranges from 0 to 100 with higher values indicating better physical functioning. The change in score, follow-up minus baseline value, ranges from -100 to +100 with higher values indicating improvement in physical functioning.
Time Frame: Baseline to 1 year
Population: Participants with both the baseline and 1 year values are included; the SF-36 was administered at a subset of clinics
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Supplemental Oxygen Therapy | No Supplemental Oxygen Therapy
Number analyzed (Participants) | 279 | 241
units on a scale | -0.5 (7.1) | -1.0 (7.4)
Statistical Analysis 1: Comparison: Supplemental Oxygen Therapy vs No Supplemental Oxygen Therapy; Test type: Superiority or Other; p = 0.71, t-test, 2 sided

9. Secondary Outcome: Sleep Quality
Description: Sleep quality is measured by the change in the Pittsburgh Sleep Quality Index total score, follow-up value minus baseline value. The Pittsburgh Sleep Quality Index total score ranges from 0 to 21 with higher values indicating worse sleep quality. The change in score, follow-up minus baseline value, ranges from -21 to +21 with higher values indicating worsening in sleep quality.
Time Frame: Baseline to 1 year
Population: Participants with both the baseline and 1 year values are included
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Supplemental Oxygen Therapy | No Supplemental Oxygen Therapy
Number analyzed (Participants) | 274 | 240
units on a scale | -0.3 (3.4) | 0.4 (3.2)
Statistical Analysis 1: Comparison: Supplemental Oxygen Therapy vs No Supplemental Oxygen Therapy; Test type: Superiority or Other; p = 0.03, t-test, 2 sided

10. Secondary Outcome: Anxiety
Description: Anxiety is measured by the change in the Hospital Anxiety and Depression Scale (HADS) anxiety score, follow-up value minus baseline value. The HADS anxiety score ranges from 0 to 21 with higher values indicating greater anxiety. The change in score, follow-up minus baseline value, ranges from -21 to +21 with higher values indicating increase in anxiety
Time Frame: Baseline to 1 year
Population: Patients with both the baseline and 1 year values are included; a subset of clinics administered the HADS questionnaire.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Supplemental Oxygen Therapy | No Supplemental Oxygen Therapy
Number analyzed (Participants) | 280 | 243
units on a scale | -0.1 (3.3) | 0.3 (3.2)
Statistical Analysis 1: Comparison: Supplemental Oxygen Therapy vs No Supplemental Oxygen Therapy; Test type: Superiority or Other; p = 0.28, t-test, 2 sided

11. Secondary Outcome: Depression
Description: Depression is measured by the change in the Hospital Anxiety and Depression Scale (HADS) depression score, follow-up value minus baseline value. The HADS depression score ranges from 0 to 21 with higher values indicating greater depression. The change in score, follow-up minus baseline value, ranges from -21 to +21 with higher values indicating increase in depression
Time Frame: Baseline to 1 year
Population: Patients with both baseline and 1 year values are included
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Supplemental Oxygen Therapy | No Supplemental Oxygen Therapy
Number analyzed (Participants) | 280 | 243
units on a scale | 0.4 (3.0) | 0.7 (2.8)
Statistical Analysis 1: Comparison: Supplemental Oxygen Therapy vs No Supplemental Oxygen Therapy; Test type: Superiority or Other; p = 0.41, t-test, 2 sided

12. Secondary Outcome: Development of Severe Resting Desaturation
Description: Severe resting desaturation is defined as resting room air SpO2 <=88%
Time Frame: Baseline to 1 year
Population: Participants completing the 1 year saturation assessment are analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | Supplemental Oxygen Therapy | No Supplemental Oxygen Therapy
Number analyzed (Participants) | 322 | 288
Participants | 7 | 3
Statistical Analysis 1: Comparison: Supplemental Oxygen Therapy vs No Supplemental Oxygen Therapy; Test type: Superiority or Other; Risk Ratio (RR) = 2.09, 95% CI 2-sided [0.54 to 8.00] — Relative risk, LTOT vs No LTOT

13. Secondary Outcome: 6-minute Walk Distance
Description: Change in distance walked during 6-minute walk test, follow-up value minus baseline value (feet)
Time Frame: Baseline to 1 year
Population: Change in 6 minute walk distance from baseline to 1 year is analyzed for patients with both baseline and 1 year values
Measure: Mean (Standard Deviation); unit: feet
Arm/Group | Supplemental Oxygen Therapy | No Supplemental Oxygen Therapy
Number analyzed (Participants) | 291 | 267
feet | -53 (281) | -85 (245)
Statistical Analysis 1: Comparison: Supplemental Oxygen Therapy vs No Supplemental Oxygen Therapy; Test type: Superiority or Other; p = 0.37, t-test, 2 sided

14. Secondary Outcome: Dyspnea
Description: Change in dyspnea is measured by change in the St George's Respiratory Questionnaire (SGRQ) total score, follow-up value minus baseline value. The SGRQ total score ranges from 0 to 100, with higher values indicating worse dyspnea. The change in score, follow-up value minus baseline value, ranges from -100 to +100, with higher values indicating increase in dyspnea.
Time Frame: Baseline to 1 year
Population: Patients with both the baseline and 1 year SGRQ total score are included
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Supplemental Oxygen Therapy | No Supplemental Oxygen Therapy
Number analyzed (Participants) | 331 | 299
units on a scale | -1.1 (13.5) | 0.6 (12.7)
Statistical Analysis 1: Comparison: Supplemental Oxygen Therapy vs No Supplemental Oxygen Therapy; Test type: Superiority or Other; p = 0.21, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Through study completion. Median follow-up of 41.5 months
Description: Adverse events reported to be possibly, probably or definitely related to use of supplemental oxygen were tracked. Mortality is reported for those assigned to Supplemental Oxygen, those assigned to No Supplemental Oxygen who crossed over to Supplemental Oxygen at some time during follow-up, and those assigned to No Supplemental Oxygen who never reported using supplemental oxygen, but we do not know whether the patient was using supplemental oxygen when death occurred.
Groups:
- Supplemental Oxygen Therapy: Participants will receive treatment with supplemental oxygen therapy. Supplemental oxygen therapy: oxygen dose at rest and during sleep will be 2 L/min via nasal cannula. The oxygen dose used while walking will be individually prescribed and will be sufficient to maintain oxygen saturation at 90% or above for at least 2 minutes while walking. Participants who have low blood oxygen levels at rest will be instructed to use oxygen 24 hours per day. Participants who have normal resting blood oxygen levels, but low or very low blood oxygen levels during exercise, will be instructed to use oxygen during physical activity and sleep.
- Patients Crossing Over to Supplemental Oxygen Therapy: Participants in the No supplemental oxygen therapy group who receive supplemental oxygen therapy during their participation in the trial due to prescription of supplemental oxygen outside the trial or development of severe resting or exercise hypoxemia
- No Supplemental Oxygen: Participants in the No supplemental oxygen who did not receive home oxygen during their participation in the trial.
Arm/Group | Supplemental Oxygen Therapy | Patients Crossing Over to Supplemental Oxygen Therapy | No Supplemental Oxygen
All-Cause Mortality (participants affected / at risk) | 66/368 | 24/125 | 49/245
Serious Adverse Events (participants affected / at risk) | 2/368 | 0/125 | 0/245
Other Adverse Events (participants affected / at risk) | 30/368 | 10/125 | 0/245
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Supplemental Oxygen Therapy (N=368) | Patients Crossing Over to Supplemental Oxygen Therapy (N=125) | No Supplemental Oxygen (N=245)
Event attributed to supplemental oxygen required hospitalization (General disorders) | 2 (2) | 0 (0) | 0 (0) — Overnight hospitalization due to injury from tripping over oxygen equipment (1 night hospitalization, humerus fracture, 1 participant; 6-day hospitalization, rib fractures, 1 participant)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Supplemental Oxygen Therapy (N=368) | Patients Crossing Over to Supplemental Oxygen Therapy (N=125) | No Supplemental Oxygen (N=245)
Fires related to oxygen use (Product Issues) | 2 (2) | 0 (0) | 0 (0) — Home fire related to oxygen use
Burn from smoking around oxygen equipment (Injury, poisoning and procedural complications) | 2 (3) | 0 (0) | 0 (0)
Burn from using oxygen equipment around open flame (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Burn from liquid oxygen frost (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 0 (0)
Nosebleed (Ear and labyrinth disorders) | 4 (4) | 4 (5) | 0 (0)
Tripping/falling over oxygen equipment not resulting in hospitalization (Injury, poisoning and procedural complications) | 13 (17) | 4 (4) | 0 (0)
Blisters on ears and ear pain (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Dry eyes (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Funny feeling in sinus area (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Increased intestinal gas (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (General disorders) | 2 (2) | 0 (0) | 0 (0)
Nausea (General disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No